CLINICAL TRIAL: NCT00662441
Title: Open-Label, Multi-Centre, Study of Levitra 10 mg Once a Day in Males With Erectile Dysfunction Was Carried Out in Four Centres Namely Lagos, Port Harcourt, Enuge and Maiduguri at Their University Teaching Hospitals
Brief Title: Evaluating of the Efficacy and Safety of Vardenafil in Subjects With Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Healthcare AG
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 100578
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 10mg taken 1 hours before sexual intercourse

SUMMARY:
Erectile dysfunction (ED) is defined as the inability to achieve or maintain an erection sufficient for satisfactory sexual performance. An ideal treatment option should be effective and reliable, have minimal side effects, be simple to use and affordable. The purpose was the evaluation of efficacy and safety of 10 mg oral Vardenafil in Nigerian subjects with Erectile Dysfunction (ED).

ELIGIBILITY:
Inclusion Criteria:

* Men >/= 18 years of age
* Erectile Dysfunction

Exclusion Criteria:

* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy
* Other exclusion criteria apply according to the Summary of Product Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-09; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
International Index of Erectile Function- Erectile Function domain | 8 weeks

SECONDARY OUTCOMES:
Global Assessment Questionnaire (GAQ) | 8 weeks
Safety and tolerability | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer